CLINICAL TRIAL: NCT04870281
Title: BIO-AffectDX Clinical Study
Brief Title: Atrial Fibrillation Associated With Heart Failure Treated by BIOTRONIK's CRT-DX System
Acronym: BIO-AffectDX
Status: Terminated | Type: Observational
Why Stopped: The study terminated due to significant delays in site start-up activities and enrollment in the setting of the ongoing COVID-19 pandemic.
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BIO-AffectDX
Record Dates: First submitted 2021-04-26; First posted 2021-05-03 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure; Atrial Fibrillation; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CRT-DX System
  Interventions: Device: CRT-DX

INTERVENTIONS:
Device: CRT-DX — Evaluation of overall health, including heart failure and atrial fibrillation improvement, changes in physical fitness, and general quality of life.

SUMMARY:
The purpose of the BIO-AffectDX Study is to prospectively evaluate improvement from baseline in heart failure subjects with atrial fibrillation (AF) implanted with a two-lead CRT-DX system, with emphasis on a comparison of patient outcomes between AF subtypes.

DETAILED DESCRIPTION:
There is a need for more evidence about the benefits of Cardiac Resynchronization Therapy (CRT) in a patient population with heart failure and atrial fibrillation. The BIO-AffectDX Study will gather information about adults with heart failure and atrial fibrillation who are treated with a CRT-DX device from many locations across the United States. The BIO-AffectDX Study will look at the results of treatment in participants with the primary goal to evaluate the improvement in overall health prior to device implant through 12 months. Overall health will be measured by your study doctor for AF improvement, physical fitness, and general quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Standard CRT-D indication according to current guidelines
* Patient has documented history of paroxysmal, persistent, or long-standing persistent atrial fibrillation
* De novo implant or upgrade from a DX implantable cardioverter-defibrillator (ICD) system
* Implant planned to occur within 30 days of consent
* Patient is able to understand English or Spanish
* Patient is able to understand the nature of the study and provide informed consent
* Patient is willing and able to complete all routine study visits at the investigational site for up to 12 months of follow-up
* Patient is willing to utilize BIOTRONIK Home Monitoring® via CardioMessenger
* Patient age is greater than or equal to 18 years

After consent has been signed, additional inclusion criteria must be fulfilled for study participation:

* Baseline subject assessment is evaluated as New York Heart Association class II, III or ambulatory IV heart failure at study Enrollment Visit
* Baseline subject assessment of six-minute walk test is completed at study Enrollment Visit and walk distance ≤ 450 meters (1,476 feet)

Exclusion Criteria:

* Contraindication to CRT-D/CRT-DX
* Patient has current or previous atrial pacing need
* Patient is considered for a His Bundle Pacing system
* Patient has current or previous pacemaker, non-DX ICD implant, or bi-ventricular pacing system prior to enrolling
* Patient is currently planned for a pulmonary vein isolation catheter ablation procedure within 3 months of consent
* Patient life expectancy is less than 1 year
* Patient is expected to receive heart transplantation or ventricular assist device within 1 year after implant
* Patient is expected to have a cardiac surgical procedure, such as coronary artery bypass graft or valve transcatheter replacement/repair or surgery, planned to occur within 6-months after implant (excludes atrioventricular node ablation procedures)
* Patient is currently on dialysis, or is expected to receive dialysis within 1 year of implant
* Patient is enrolled in any investigational cardiac device or drug trial that might significantly affect the studied outcomes
* Any condition (e.g. severe arthritis, wheelchair bound, etc.) preventing the patient from performing the required six-minute walk test
* Conditions that prohibit placement of any of the system leads
* Patient reports pregnancy at the time of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients selected for participation should be from the investigator's general patient population with standard CRT-D indication and according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Composite Score from baseline | 12 months

SECONDARY OUTCOMES:
Rate of composite all-cause death and heart failure | 12 months
Change in quality of life questionnaires from baseline for all patients and by atrial fibrillation sub-type | 6 and 12 months
Change in New York Heart Association class from baseline for all patients and by atrial fibrillation sub-type | 6 and 12 months
Change in six-minute walk distance from baseline for all patients and by atrial fibrillation sub-type | 6 and 12 months
Change in atrial fibrillation burden from baseline for all patients and by atrial fibrillation sub-type | 6 and 12 months
Change in Clinical Composite Score from baseline | 6 months
Rate of major complications | 12 months
Rate of conversion to sinus rhythm | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Costea, MD, Study Chair — University of Cincinnati Heart
Locations (23):
- United States (23):
  - University of California San Diego - La Jolla, La Jolla, California
  - Cardiology Associates Medical Group, Ventura, California
  - Orlando Health Heart Institute, Orlando, Florida
  - AdventHealth Tampa, Tampa, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky - Gill Heart and Vascular Institute, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - Mercy Hospital Springfield, Springfield, Missouri
  - Glacier View Research Institute Cardiology, Kalispell, Montana
  - Weill Cornell Medicine, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Heart Rhythm Associates, Greenville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - ProMedica Northwest Ohio Cardiology Consultants, Toledo, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Upstate Cardiology, Greenville, South Carolina
  - Erlanger Institute for Clinical Research, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Applicable de-identified individual participant data will be made available to achieve aims in approved proposals, including but not limited to sub-analysis or meta-analysis that are not specifically pre-planned within the protocol.
Supporting Information: Study Protocol
Time Frame: Beginning no later than 12 months and ending no earlier than 3 years following study closure.
Access Criteria: Proposals should be directed to BIOTRONIK Clinical Studies (BIOTRONIK Inc., Attn: Clinical Studies, 6024 Jean Road, Lake Oswego, OR 97035; 1-800-547-0394). BIOTRONIK, in consultation with the BIO-AffectDX Steering Committee, will review and evaluate proposals for scientific merit, fiscal feasibility, and logistical feasibility. They will additionally consider if the proposed publication fits into the overall BIO-AffectDX publication plan. If approved, the data requestors will need to sign a data use/access agreement prior to obtaining the data and agree to review and input from the BIO-AffectDX Steering Committee members.